CLINICAL TRIAL: NCT04529967
Title: Child-Parent Screening of Familial Hypercholesterolemia in Children
Brief Title: Child-Parent Familial Hypercholesterolemia Screening
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: CHFD-2020007
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — capillary blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no interventions — it is a observational study, do not have interventions.

SUMMARY:
Child-parent screening for familial hypercholesterolemia has been proposed to identify children and their parent who are carrier of mutations and with high risk for inherited premature coronary artery disease. The investigators assessed the efficacy and feasibility of such screening in primary care practice.

key scientific questions:

1. The 95th and 99th percentile of finger blood TC in children of 2 years old.
2. Mutations that contribute to high TC status ( serum TC >99th percentiles) compared with international FH48 panel for FH genetic screening.

DETAILED DESCRIPTION:
Familial hypercholesterolemia (FH) is an inherited condition resulting in high levels of low-density lipoprotein cholesterol (LDL-C) and increased risk of premature coronary artery disease in men and women. Child-parent screening for familial hypercholesterolemia has been proposed to identify persons who are carriers of FH mutations and with high risk for inherited premature coronary artery disease. The investigators will conduct a cross-sectional community-based screening in children of 2 years old to detect FH children cases using finger blood TC test first and followed by serum TC test and mutation test, and to identify and diagnose their affected parents. This study aims to established the child-parent screening program and technique issues for early diagnosis of familial hypercholesterolemia families for future early intervention.

Child-parent screening strategy in our study consists three steps: i. Capillary blood total cholesterol test of children aged around 2 years; ii. re-test for children with cholesterol>95th percentile in the first step; iii. WES (whole exome sequencing) test for >P99 in the first two steps. iV: TC test and mutation test to the parents of the child FH cases. The investigators will determine FH families based on the program. Children's Hospital of Fudan University will provide treatment further.

ELIGIBILITY:
Inclusion Criteria:

* Receive routine child care
* aged 1 - 3 years old ( date of investigate minus date of birth)

Exclusion Criteria:

* It is up to the researcher to decide whether it is suitable to participate in this research

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All community-children from slelected communities aged 1 to 3 who receive regular child care (programmed immunization vaccination clinic) within a prespecified study period
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The affected status of Familial Hypercholesterolemia | At enrollment
  heterozygote or homozygote carriers of established FH mutations in LDLR, PSCK9 and APOB gene, including mutations included in the FH48 and new ones identified in Chinese children

SECONDARY OUTCOMES:
fasting total cholesterol level by Fingertip capillary blood test in children around 2 years old | At enrollment
affected status of known FH mutation | At enrollment
  according to FH48
fasting serum LDL-c levels of children with finger TC over P95 | At enrollment

CONTACTS AND LOCATIONS:
Overall Officials: LIling Qian, Master, Study Director — Children's Hospital of Fudan University; Rui Dong, MD, Study Director — Children's Hospital of Fudan University
Locations (6):
- China (6):
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - Qidong Women and Children Hospital, Qidong, Jiangsu
  - Weili Yan, Shanghai, Shanghai Municipality
  - Shanxi Provincial Children's Hospital, Taiyuan, Shanxi
  - Chongqin Medical University Affiliated Children's Hospital, Chongqing, Sichuan
  - Urumqi Children's Hospital, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: Undecided
The data generated and/or during current study are not publicly available due to incomplete study, but are available from the corresponding author on reasonable request.